CLINICAL TRIAL: NCT05069675
Title: Incidence and Risk Factors for Cystoid Macular Edema After Primary Vitrectomy With Gas Tamponade for Rhegmatogenous Retinal Detachment: a National Study Group
Brief Title: Cystoid Macular Edema After Vitrectomy for Rhegmatogenous Retinal Detachment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Antonio Longo, Associate Professor, University of Catania
Other Study IDs: 69/2021/PO
Record Dates: First submitted 2021-09-20; First posted 2021-10-06 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Cystoid Macular Edema
Keywords: cystoid macular edema; rhegmatogenous retinal detachment; vitrectomy; gas tamponade
MeSH Terms: conditions — Macular Edema | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vitrectomy — vitrectomy with gas tamponade

SUMMARY:
To investigate the incidence of cystoid macular edema in eyes with primary rhegmatogenous retinal detachment successfully treated with vitrectomy with gas tamponade, and to evaluate the clinical variables associated with its development.

DETAILED DESCRIPTION:
this is an observational, retrospective, multicentre study. The study is based on the retrospective collection of clinical data from patients undergoing gas tamponade vitrectomy for rhegmatogenous retinal detachment. The collection of such data by the investigators will take place at each participating center anonymously.

demographics, systemic, and preoperative, intraoperative and post-operative data will be collected The sample size was calculated to obtain approximately 200 patients with cystoid macular edema. Since cystoid macular edema has been detected in 13% of patients after retinal detachment gas vitrectomy, and assuming that this event can occur between 10% and 15% of cases, the study will include at least 2000 cases.

ELIGIBILITY:
Inclusion Criteria:

* primary rhegmatogenous retinal detachment treated with vitrectomy with gas tamponade;
* follow-up of 3 months or more;
* age > 18 years ;
* no previous eye surgery, except cataract surgery performed at least 6 months after hospitalization for retinal detachment;
* anatomical success, i.e. retinal re-attachment, after a single gas vitrectomy;
* no other eye surgery during follow-up;
* availability of optical coherence tomography (OCT) imaging

Exclusion Criteria:

* history of other eye diseases (glaucoma, age-related macular degeneration, uveitis, diabetic retinopathy, maculopathy);
* macular hole;
* recurrent retinal detachment;
* use of silicone oil is used as a tamponading agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with primary regmatogenous retinal detechment successfully treated by vitrectomy with gas tamnponade at several Eye Centers, will be included in the study.
  clinical data will be retrospectively retrieved.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
incidence of cystoid macular edema | from 1 month up to 6 months after surgery
  cystoid macular edema assessed by OCT (central subfield thickness >310 micron, with presence of intraretinal cystic areas of low reflectivity in OPL) visual acuity

SECONDARY OUTCOMES:
factors related to development of macular edema | from 1 month up to 6 months after surgery
  demographics, systemic and ocular parameters

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Eye Clinic, University of Bari, Bari
  - Eye Clinic, Humanitas University, Bergamo
  - Eye Clinic, Azienda Policlinico San Marco, Catania
  - Eye Clinic, University of Palermo, Palermo
  - Eye Clinic, University of Perugia, Perugia
  - Eye Clinic University of Turin, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatziralli I, Theodossiadis G, Dimitriou E, Kazantzis D, Theodossiadis P. Macular Edema after Successful Pars Plana Vitrectomy for Rhegmatogenous Retinal Detachment: Factors Affecting Edema Development and Considerations for Treatment. Ocul Immunol Inflamm. 2021 Jan 2;29(1):187-192. doi: 10.1080/09273948.2019.1652330. Epub 2019 Oct 2. PMID 31577459
- [Background] Banker TP, Reilly GS, Jalaj S, Weichel ED. Epiretinal membrane and cystoid macular edema after retinal detachment repair with small-gauge pars plana vitrectomy. Eur J Ophthalmol. 2015 Nov-Dec;25(6):565-70. doi: 10.5301/ejo.5000609. Epub 2015 Apr 15. PMID 25907288
- [Background] Joseph DP, Ryan EH, Ryan CM, Forbes NJK, Wagley S, Yonekawa Y, Mittra RA, Parke DW, Emerson GG, Shah GK, Blinder KJ, Capone A, Williams GA, Eliott D, Gupta OP, Hsu J, Regillo CD. Primary Retinal Detachment Outcomes Study: Pseudophakic Retinal Detachment Outcomes: Primary Retinal Detachment Outcomes Study Report Number 3. Ophthalmology. 2020 Nov;127(11):1507-1514. doi: 10.1016/j.ophtha.2020.05.005. Epub 2020 May 8. PMID 32437865